CLINICAL TRIAL: NCT03477344
Title: Dexmedetomidine After Cardiac Surgery for Prevention of Delirium: The Exactum Study a Randomised Double Blind Controlled Trial
Brief Title: Dexmedetomidine After Cardiac Surgery for Prevention of Delirium
Acronym: EXACTUM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Collaborators: Direction Générale de l'Offre de Soins (Other Government); Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 29BRC18.0051 (EXACTUM)
Record Dates: First submitted 2018-03-06; First posted 2018-03-26 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: ICU Delirium
Keywords: Cardiac Surgery; Delirium; Sleep deprivation
MeSH Terms: conditions — Delirium; Sleep Deprivation | interventions — Dexmedetomidine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmédétomidine (Active Comparator): Intravenous infusion with electric syringe of Dexmedetomidine 0,4ug/ml. Rate 0,1ug/kg/h to 1,4ug/kg/h. Nightly infusion from 20:00 to 08:00. The drug is titrated to achieve RASS between -1 and 1. Modification of infusion rate by 0,1ug/kg/h is recommended with stabilization phase of 1 hour before another rate adjustment.
  Interventions: Drug: Dexmedetomidine
- Sodium Chloride 0,9% (Placebo Comparator): Intravenous infusion with electric syringe of normal saline. Rate modifications follow the same rules as in experimental group.
  Interventions: Drug: Sodium chloride 0.9%

INTERVENTIONS:
Drug: Dexmedetomidine — Intravenous infusion with electric syringe of Dexmedetomidine 0,4ug/ml. Rate 0,1ug/kg/h to 1,4ug/kg/h. Nightly infusion from 20:00 to 08:00. The drug is titrated to achieve RASS between -1 and 1. Modification of infusion rate by 0,1ug/kg/h is recommended with stabilization phase of 1 hour before another rate adjustment.
  Arms: Dexmédétomidine
Drug: Sodium chloride 0.9% — Intravenous infusion with electric syringe of normal saline. Rate modifications follow the same rules as in experimental group.
  Arms: Sodium Chloride 0,9%

SUMMARY:
We designed a prospective, double blind, randomized, controlled versus placebo study to evaluate the efficacy of nightly low dose of Dexmedetomidine infusion to promote sleep and lower delirium in a population of post cardiac surgery patients. This population is characterized by longer ICU stay, more physical restraints such as catheters and drains, pain and sleep deprivation. It is associated with higher prevalence of Delirium and agitation leading to exposure to severe agitation related adverse events.

DETAILED DESCRIPTION:
Delirium occurs in about 25% of patients after cardiac surgery. It is an independent factor of poor outcome and recovery after ICU stay as it is associated with mortality and impaired mental function one year after its onset. It is associated with increased public health costs during the hospital stay and after.

The use of Dexmedetomidine as sedative medication is more and more described. It is well established that it can lower delirium onset comparatively to Midazolam or Propofol. It is also useful in agitated delirium as a complementary medication to reduce delirium duration. A study published by Su et al in 2016 assessed the efficacy of Dexmedetomidine in prevention of post-surgical delirium for patients older than 65 years after non cardiac surgery. Patients were mainly admitted in the ICU after abdominal surgery for malignant tumor. Dexmedetomidine was used at very low dose to promote sleep during ICU stay. In this study the onset of delirium was significantly lowered by one half for the first week after surgery. However, this study only focused on older patients and non-cardiac surgery population with short mechanical ventilation duration, short ICU stay and low incidence of complications.

We designed a prospective, double blind, randomized, controlled versus placebo study to evaluate the efficacy of nightly low dose of Dexmedetomidine infusion to promote sleep and lower delirium in a population of post cardiac surgery patients. This population is characterized by longer ICU stay, more physical restraints such as catheters and drains, pain and sleep deprivation. It is associated with higher prevalence of Delirium and agitation leading to exposure to severe agitation related adverse events. In the study by Su and al low dose Dexmedetomidine did not induce adverse events such as bradycardia or hypotension, conversely safety outcomes showed that Dexmedetomidine use was associated with fewer tachycardia and hypoxaemia. Moreover, data shows that Dexmedetomidine is likely to play a cardio protective role in the same way as Clonidine. Those findings are encouraging for its use after cardiac surgery.

Delirium will be assessed by the Confusion Assessment Method for the ICU (CAM ICU) and the primary endpoint of the study is the occurrence of delirium in the first 7 days following surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 65 or more who undergo cardiac surgery on and off-pump: coronary artery bypass graft, cardiac valve replacement or both.
* Consent signed

Exclusion Criteria:

* history of mental illness, dementia
* inclusion in another study evaluating sedation or pain
* length of stay in ICU less than 24 hours
* alpha 2 agonists allergy
* surgery performed in an immediate emergency situation
* uncontrolled hypotension
* second and third degree atrioventricular block without pacemaker
* severe hepatic insufficiency
* acute cerebrovascular diseases
* patient treated with clonidine
* patient with disturbed preoperative liver assessment (hepatocellular insufficiency)
* patient under guardianship or curatorship

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 348 (Actual)
Dates: Start 2019-01-04 (Actual); Primary Completion 2021-06-29 (Actual); Study Completion 2021-06-29 (Actual)

PRIMARY OUTCOMES:
Delirium | 7 days
  Occurrence of delirium diagnosed by the Confusion Assessment Method (CAM ICU) at any time in the first seven days after surgery

SECONDARY OUTCOMES:
agitation with be assessed using the Richmond agitation and sedation score | 7 days
  Score Term Description
  * 4 Combative Overtly combative or violent; immediate danger to staff
  * 3 Very agitated Pulls on or removes tube(s) or catheter(s) or has aggressive behavior toward staff
  * 2 Agitated Frequent nonpurposeful movement or patient-ventilator dyssynchrony
  * 1 Restless Anxious or apprehensive but movements not aggressive or vigorous 0 Alert and calm Spontaneously pays attention to caregiver
    * 1 Drowsy Not fully alert, but has sustained (more than 10 seconds) awakening, with eye contact, to voice
    * 2 Light sedation Briefly (less than 10 seconds) awakens with eye contact to voice
    * 3 Moderate sedation Any movement (but no eye contact) to voice
    * 4 Deep sedation No response to voice, but any movement to physical stimulation
    * 5 Unarousable No response to voice or physical stimulation
length of ICU stay | 28 days
  Lenght of patient's ICU stay
length of hospital stay | 28 days
  Length of Patient's hospital stay
quality of life 3 months after surgery with the The Short Form (36) Health Survey score | 90 days
  The Short Form (36) Health Survey is a 36-item, patient-reported survey of patient health. The SF-36 is a measure of health status and an abbreviated variant of it, the SF-6D, is commonly used in health economics as a variable in the quality-adjusted life year calculation to determine the cost-effectiveness of a health treatment. The original SF-36 came out from the Medical Outcome Study, MOS, done by the RAND Corporation. Since then a group of researchers from the original study released a commercial version of SF-36 while the original SF-36 is available in public domain license free from RAND.
cognitive capacity 3 months after surgery evaluated with the Cognitive Failures Questionnnaire (CFQ) | 90 days
  The Cognitive Failures Questionnaire is a self-report scale that taps failures in everyday actions, perception and attention, and memory over the last month. It consists of 25 items that are scored on a 5-point scale (0=never; 4=very often). Illustrative items are 'Do you fail to notice signposts on the road?' and 'Do you forget where you put something like a newspaper or a book?' Scores are summed to obtain a total CFQ score varying from 0 to 100, with higher scores indicating more self-reported cognitive failures.
agitation related adverse events onset and number | 7 days
  -self-extubation
agitation related adverse events onset and number | 7 days
  -catheter or medical devices removal (drains, urinary catheter, arterial and central venous catheters, externenal pacemaker)
agitation related adverse events onset and number | 7 days
  -fall of bed
agitation related adverse events onset and number | 7 days
  -getaway
agitation related adverse events onset and number | 7 days
  -contention removal
agitation related adverse events onset and number | 7 days
  -aggressive acts
Self-assessment of sleep quality | 7 days
  Assessment by a numerical scale from 0 to 10 and the Leeds Sleep questionnaire
Intra hospital mortality and Mortality at 3 months of surgery | 3 months
Cognitive capacity | 3 months
  Cognitive capacity assessed by Cognitive Failures Questionnaire (CFQ) at 3 months of surgery
Post-traumatic stress disorder | 3 months
  Post-traumatic stress disorder assessed by the PCL-5 questionnaire at 3 months of surgery

CONTACTS AND LOCATIONS:
Locations (9):
- France (9):
  - Angers university hospital, Angers
  - CHRU de Brest, Brest
  - Clermont Ferrand university hospital, Clermont-Ferrand
  - CHU de Grenoble, Grenoble
  - Hôpital Privé Jacques Cartier, Massy
  - CHU de Nantes, Nantes
  - CHU la Pitié Salpétrière, Paris
  - CHU Poitiers, Poitiers
  - CHU de Rennes, Rennes

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning five years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.

REFERENCES:
- [Derived] Huet O, Gargadennec T, Oilleau JF, Rozec B, Nesseler N, Bougle A, Kerforne T, Lasocki S, Eljezi V, Dessertaine G, Amour J, Chapalain X; EXACTUM and the Atlanrea Study Group. Prevention of post-operative delirium using an overnight infusion of dexmedetomidine in patients undergoing cardiac surgery: a pragmatic, randomized, double-blind, placebo-controlled trial. Crit Care. 2024 Feb 29;28(1):64. doi: 10.1186/s13054-024-04842-1. PMID 38419119
- [Derived] Gargadennec T, Oilleau JF, Rozec B, Nesseler N, Lasocki S, Futier E, Amour J, Durand M, Bougle A, Kerforne T, Consigny M, Eddi D, Huet O. Dexmedetomidine after Cardiac Surgery for Prevention of Delirium (EXACTUM) trial protocol: a multicentre randomised, double-blind, placebo-controlled trial. BMJ Open. 2022 Apr 8;12(4):e058968. doi: 10.1136/bmjopen-2021-058968. PMID 35396310